CLINICAL TRIAL: NCT04061733
Title: New Hydroxyethyl Cellulose Hydrogel for the Treatment of the Pain of Knee Arthrosis
Acronym: PROMGEL-OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Promedon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMGEL-OA-2018
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: osteoarthritis; pain; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Subjects who will receive an injection of the hydrogel
  Interventions: Device: Hydrogel injection

INTERVENTIONS:
Device: Hydrogel injection — Hydrogel injection

SUMMARY:
Prospective, multicenter study, unmasked, single-arm, to study the safety and efficacy of a new hydroxyethyl cellulose hydrogel for the treatment of the knee pain caused by osteoarthritis.

DETAILED DESCRIPTION:
Prospective, multicenter study, unmasked, single-arm, to study the safety and efficacy of a new hydroxyethyl cellulose hydrogel for the treatment of the knee pain caused by osteoarthritis. The working hypothesis is that the effect of hydrogel use on the study population will result in a reduction in pain in the knees affected by symptomatic OA.

The general objective of this study is to generate clinical evidence of the safety and efficacy of the new hydrogel used as a treatment of symptomatic knee osteoarthritis.

The patient's perception of the pain caused by osteoarthritis in the knee joint before and after the treatment under evaluation will be quantify. Subjects' quality of life before and after treatment will also be evaluated. Monitoring of the adverse events associated with the use of the device under evaluation will be determined. Subjects will be follow-up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with osteoarthritis of unilateral or bilateral knee osteoarthritis who meet the criteria defined by the American College of Rheumatology for at least 4 months prior to the study. In bilateral knee osteoarthritis, only the knee with more symptoms will be treated.
2. Arthrosis grade 2 or 3 according to the Kellgren - Lawrence Classification System (radiological classification)
3. Persistence of symptoms despite conservative treatment (NSAIDS, Physical Therapy, lifestyle changes, etc.) for more than 4 months
4. Subjects aged between 40 and 70 years
5. BMI (Kg/m²) 20-32
6. For female subjects: postmenopausal women with at least 1 year documented in the medical record.

Exclusion Criteria:

1. Arthrosis grade 0 or 4 according to the Kellgren - Lawrence Classification
2. History of allergy to any of the Hydrogel components
3. History of previous treatment with corticosteroid injections less than 4 months prior to entry into this clinical study
4. History of previous treatment with hyaluronic acid viscosupplementation
5. History of open or arthroscopic surgery in the knee to be treated less than 9 months
6. Severe chronic progressive disease
7. Insulin-requiring diabetes
8. Rheumatic diseases (rheumatoid arthritis, psoriasis, gout, pseudo-gout, fibromyalgia)
9. History of septic arthritis
10. History of psychiatric illness that makes it impossible to understand and sign the informed consent
11. History or presence of severe peripheral vascular disease
12. Deseje over 15° valgus or varus movement
13. Pregnant or breastfeeding women
14. BMI (kg/m²)> 32

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain assessment: Percentage of pain reduction using a visual analogue scale | Change from Baseline at postoperative 12 months follow-up
  Percentage of pain reduction using a visual analogue scale (Wong-Baker scale) where Face 0: does not hurt at all and Face 10: hurts as much as you can imagine

SECONDARY OUTCOMES:
Improvement of Quality of life: KOOS | Baseline, and postoperative at 1, 3, 6 and 12 months follow-up
  Quality of life (QoL-Status) - defined as improvement of the QoL of the subjects, compared to the baseline values for KOOS (Knee injury and Osteoarthritis Outcome Score) questionnaire.
  The KOOS questionnaire was developed as an instrument to assess the patient's opinion about their knee and associated problems.The KOOS questionnaire measures 5 subscales: pain referred by the patient, other specific symptoms of the disease, function in daily life activities, function in sport and recreation and quality of life related to the knee. All items have 5 possible response options (from 0 to 4) where 0 indicates no problems and 4 indicates extreme problems, and each of those 5 scores is calculated as the sum of the included items. The scores are transformed on a scale of 0 to 100, which 0 represents extreme knee problems and 100 indicates no symptoms. The score ranges from 0 to 100, separately for each sub-scale. A change of 10 points or more is considered a clinically significant change.
Improvement of Health status | Change from Baseline at postoperative at 1, 3, 6 and 12 months follow-up
  Health Status assessed with 12-Item Short-Form Health Survey (SF-12). It consists of 12 items (grouped in 8 health concepts: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health) from which two summaries are constructed: physical and mental. The higher the score on the scales indicates the better health.
Patient Global Impression | Change from Baseline, up to three days after injection, postoperative at 1, 3, 6 and 12 months follow-up
  Patient Global Impression with the his/her osteoarthritis will be evaluated with a visual analogue scale (Wong-Baker scale) where Face 0: represents an inactive osteoarthritis, that is, without symptoms and Face 10: represents a very active osteoarthritis, that is, with severe symptoms.
Rate of Adverse Events | At injection, at three days after injection, postoperative at 1, 3, 6 and 12 months follow-up
  All adverse events will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando E. Barclay, Dr., Principal Investigator — IADT
Locations (3):
- Argentina (3):
  - CEMIC, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
  - IADT, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] McAlindon T, Dieppe P. Osteoarthritis: definitions and criteria. Ann Rheum Dis. 1989 Jul;48(7):531-2. doi: 10.1136/ard.48.7.531. No abstract available. PMID 2673078
- [Background] Bijlsma JW, Berenbaum F, Lafeber FP. Osteoarthritis: an update with relevance for clinical practice. Lancet. 2011 Jun 18;377(9783):2115-26. doi: 10.1016/S0140-6736(11)60243-2. PMID 21684382
- [Background] Zhang W, Doherty M, Peat G, Bierma-Zeinstra MA, Arden NK, Bresnihan B, Herrero-Beaumont G, Kirschner S, Leeb BF, Lohmander LS, Mazieres B, Pavelka K, Punzi L, So AK, Tuncer T, Watt I, Bijlsma JW. EULAR evidence-based recommendations for the diagnosis of knee osteoarthritis. Ann Rheum Dis. 2010 Mar;69(3):483-9. doi: 10.1136/ard.2009.113100. Epub 2009 Sep 17. PMID 19762361
- [Background] Bellamy N, Campbell J, Robinson V, Gee T, Bourne R, Wells G. Viscosupplementation for the treatment of osteoarthritis of the knee. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD005321. doi: 10.1002/14651858.CD005321.pub2. PMID 16625635
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Johnson VL, Hunter DJ. The epidemiology of osteoarthritis. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):5-15. doi: 10.1016/j.berh.2014.01.004. PMID 24792942
- [Background] Allen KD, Golightly YM. State of the evidence. Curr Opin Rheumatol. 2015 May;27(3):276-83. doi: 10.1097/BOR.0000000000000161. PMID 25775186
- [Background] Hunter DJ. Viscosupplementation for Osteoarthritis of the Knee. N Engl J Med. 2015 Jun 25;372(26):2570. doi: 10.1056/NEJMc1505801. No abstract available. PMID 26107064
- [Background] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- [Background] Oliveria SA, Felson DT, Reed JI, Cirillo PA, Walker AM. Incidence of symptomatic hand, hip, and knee osteoarthritis among patients in a health maintenance organization. Arthritis Rheum. 1995 Aug;38(8):1134-41. doi: 10.1002/art.1780380817. PMID 7639811
- [Background] Plotnikoff R, Karunamuni N, Lytvyak E, Penfold C, Schopflocher D, Imayama I, Johnson ST, Raine K. Osteoarthritis prevalence and modifiable factors: a population study. BMC Public Health. 2015 Nov 30;15:1195. doi: 10.1186/s12889-015-2529-0. PMID 26619838
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774
- [Background] Jevsevar DS, Brown GA, Jones DL, Matzkin EG, Manner PA, Mooar P, Schousboe JT, Stovitz S, Sanders JO, Bozic KJ, Goldberg MJ, Martin WR 3rd, Cummins DS, Donnelly P, Woznica A, Gross L; American Academy of Orthopaedic Surgeons. The American Academy of Orthopaedic Surgeons evidence-based guideline on: treatment of osteoarthritis of the knee, 2nd edition. J Bone Joint Surg Am. 2013 Oct 16;95(20):1885-6. doi: 10.2106/00004623-201310160-00010. No abstract available. PMID 24288804
- [Background] Strand V, McIntyre LF, Beach WR, Miller LE, Block JE. Safety and efficacy of US-approved viscosupplements for knee osteoarthritis: a systematic review and meta-analysis of randomized, saline-controlled trials. J Pain Res. 2015 May 7;8:217-28. doi: 10.2147/JPR.S83076. eCollection 2015. PMID 26005358
- [Background] Pal S, Thuppal S, Reddy KJ, Avasthi S, Aggarwal A, Bansal H, Mohanasundaram S, Bailleul F. Long-Term (1-Year) Safety and Efficacy of a Single 6-mL Injection of Hylan G-F 20 in Indian Patients with Symptomatic Knee Osteoarthritis. Open Rheumatol J. 2014 Oct 2;8:54-68. doi: 10.2174/1874312901408010054. eCollection 2014. PMID 25328555
- [Background] Chevalier X, Jerosch J, Goupille P, van Dijk N, Luyten FP, Scott DL, Bailleul F, Pavelka K. Single, intra-articular treatment with 6 ml hylan G-F 20 in patients with symptomatic primary osteoarthritis of the knee: a randomised, multicentre, double-blind, placebo controlled trial. Ann Rheum Dis. 2010 Jan;69(1):113-9. doi: 10.1136/ard.2008.094623. PMID 19304567
- [Background] Berenbaum F, Grifka J, Cazzaniga S, D'Amato M, Giacovelli G, Chevalier X, Rannou F, Rovati LC, Maheu E. A randomised, double-blind, controlled trial comparing two intra-articular hyaluronic acid preparations differing by their molecular weight in symptomatic knee osteoarthritis. Ann Rheum Dis. 2012 Sep;71(9):1454-60. doi: 10.1136/annrheumdis-2011-200972. Epub 2012 Jan 31. PMID 22294639
- [Background] Evaniew N, Simunovic N, Karlsson J. Cochrane in CORR(R): Viscosupplementation for the treatment of osteoarthritis of the knee. Clin Orthop Relat Res. 2014 Jul;472(7):2028-34. doi: 10.1007/s11999-013-3378-8. Epub 2013 Nov 12. No abstract available. PMID 24218162
- [Background] Campbell J, Bellamy N, Gee T. Differences between systematic reviews/meta-analyses of hyaluronic acid/hyaluronan/hylan in osteoarthritis of the knee. Osteoarthritis Cartilage. 2007 Dec;15(12):1424-36. doi: 10.1016/j.joca.2007.01.022. Epub 2007 Apr 19. PMID 17448701
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Rutjes AW, Juni P, da Costa BR, Trelle S, Nuesch E, Reichenbach S. Viscosupplementation for osteoarthritis of the knee: a systematic review and meta-analysis. Ann Intern Med. 2012 Aug 7;157(3):180-91. doi: 10.7326/0003-4819-157-3-201208070-00473. PMID 22868835
- [Background] Vaquero J, Longo UG, Forriol F, Martinelli N, Vethencourt R, Denaro V. Reliability, validity and responsiveness of the Spanish version of the Knee Injury and Osteoarthritis Outcome Score (KOOS) in patients with chondral lesion of the knee. Knee Surg Sports Traumatol Arthrosc. 2014 Jan;22(1):104-8. doi: 10.1007/s00167-012-2290-1. Epub 2012 Nov 10. PMID 23143387